CLINICAL TRIAL: NCT06401304
Title: Oncologic, Cosmetic and Patient Reported Outcomes in Value-Based Breast Surgery. A Multicentre, Cohort Study
Brief Title: Oncologic, Cosmetic and Patient Reported Outcomes in Value-Based Breast Surgery (OnCoPRO Value)
Acronym: OncoPROValue-1
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); Royal Marsden NHS Foundation Trust (Other); Westmead Breast Cancer Institute, Sydney University, Sydney, Australia (Unknown); Breast Unit, University Campus Biomedico, Rome, Italy (Unknown)
Responsible Party: Principal Investigator, Andreas Karakatsanis, Associate Professor, MD, PhD, Uppsala University
Other Study IDs: UUBreast04
Record Dates: First submitted 2024-04-27; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Breast Carcinoma in Situ; Breast Cancer Invasive; Breast Asymmetry
Keywords: Oncoplastic breast conservation; Breast Conserving Surgery; Patient reported outcomes; Shared decision making
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Anisomastia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aspires to provide outcomes on surgery, quality of life and time-to-event outcomes following the development and validation of a standardised surgical assessment tool in a shared decision-making framework for patients with pre-invasive or invasive breast cancer with breast conservation.

DETAILED DESCRIPTION:
Oncoplastic breast-conserving surgery (OPBCS) has gained increasing popularity over the last years and tends to be considered the standard of care in surgical practice. OPBCS allows for the resection of larger volumes and tumors with acceptable cosmesis, by incorporating different techniques that have evolved mainly from mastopexy, mammoplasty, and breast reduction or volume replacement techniques, such as perforator flap reconstruction.

However, no randomized controlled trial data on indications, methods, decision-making and outcomes are available, and present practice is largely based on evidence from cohort data derived from single- or multi-institutional series. Along with that, the fact that surgical decision-making in OPBCS is highly individualized renders any effort for standardization of these operations highly challenging and controversial. This is a multifactorial phenomenon, owing to anatomic differences such as breast volume, breast shape, lesion volume, localization, ptosis, body mass index (BMI) but also patient preference and availability of surgical techniques. Efforts for standardization of techniques based on tumor location, breast size, and ptosis have been made, but they do not address the principle of tailored treatment and do not cover all clinical scenarios.

On the other hand, breast-conserving surgery (BCS) followed by whole breast irradiation (WBI) yields comparable to better outcomes compared with mastectomy without WBI in terms of survival, but much better in terms of quality of life (QoL) and patient-reported outcomes and measures (PROMS), even when compared to the reconstructed breast. At the same time, OPBCS seems to yield superior cosmesis and patient satisfaction compared to traditional wide local excisions (WLE), but it is unclear whether this comes at the cost of increased morbidity or unnecessary revisionary procedures, with an impact on the delivery of systemic treatment, QoL and health economy. In addition, patient preference is a factor that precludes randomization to the method of operation in the traditional meaning, as it would not be ethical to randomize surgery that may be unnecessarily extensive or oncologically dubious. Moreover, surgeon and patient preferences and expectations may involve bias which is hard to define and a non-randomized study on the subject of WLE vs OPBCS could inevitably be unclear in how to address this inherent flaw.

PROMS such as QoL and cosmesis are even more important in the case of benign lesions that need to be operated on. This has to do with the fact that no compromises need to be made for the sake of a radical breast cancer operation as well as that benign breast surgery is more common in women of younger age. There, despite the instinctive assessment that a well-placed incision should have better outcomes, there is a complete lack of high-quality data on the matter.

At the same time, the decision-making process of the choice of surgical technique is a phenomenon poorly investigated; surgeons tend to offer the techniques they are most comfortable with and offer therapy per patient preference largely dependent on the health setting. This may account for the lack of consistency in identifying factors related to re-excision, postoperative complications, and PROMS. In this procedure, patient preference has shown to vary depending on surgical consultation, not only on the choice not to undergo mastectomy but also on the extent of BCS. Another fact that needs to be taken into account is that, despite that several classification systems and algorithms have been proposed, everyday clinical practice represents more of a continuum. On the other hand, "standard surgical assessment" performed by breast surgeons is likely to reflect personal preferences, techniques one may be most comfortable with as well as variances in healthcare provision.

This may account for the lack of consistency in practice, resulting either in involved margins and requiring re-excision, with consequences on cosmesis and patient satisfaction (undertreatment), or the unnecessary utilization of OPBCS in cases where "simpler" could produce equivalent results with less operative time, complications or need for contralateral symmetrization (overtreatment). Therefore, any objective associations between the method of BCS and outcomes remain to be elucidated.

The rationale is to investigate whether the development of a tool for surgical decision-making may facilitate the identification of appropriate surgical techniques for each patient.

The trial aims to investigate whether the application of a structured approach to select an appropriate surgical technique may have an impact on PROMS, complications, QoL, and health-economy. In that way, the effect of rationalized versus empiric employment of operative techniques (OPBCS vs WLE) may be elucidated. Additionally, it will allow for the accumulation of evidence regarding OPBCS in a way that does not come in conflict with ethics, patient preference, and real-world clinical practice. Moreover, the study will aspire to investigate whether there may be a more objective manner to define the minimum required type of surgery to obtain clear margins whilst maintaining breast function and form in a manner compatible with patient preference and optimal quality of life. As this is a multifaceted question, it is appropriate to examine it separately for different subgroups (volume replacement or displacement). Last but not least, the study may help elucidate the impact of locoregional and systemic oncologic treatment (radiotherapy, local and/or locoregional, and chemotherapy, immunotherapy, and endocrine therapy) in PROMS on the type of surgical treatment the patient has received. The design is intended to be highly pragmatic. Therefore, the systematic restructuring and the capitalization of the routinely available preoperative patient data will be used towards the effort of developing a clinical decision-making tool.

The study will look into surgical outcomes (complications, re-excision rates, conversion to mastectomy), patient-reported outcomes and experience, time-to-event outcomes (local recurrence-free survival, locoregional recurrence-free survival, disease-free survival, and overall survival) as well as health economy factors. These will be examined on an individual participant level, and a subgroup level, such as per oncoplastic reconstructive principle (volume displacement vs volume replacement), different oncoplastic techniques (eg. mastopexies vs reduction vs perforator flaps), onco-cosmetic surgery or not, concomitant contralateral symmetrization or not.

Oncoplastic breast-conserving surgery (OPBCS) has gained increasing popularity over the last years and tends to be considered the standard of care in surgical practice. OPBCS allows for the resection of larger volumes and tumors with acceptable cosmesis, by incorporating different techniques that have evolved mainly from mastopexy, mammoplasty, and breast reduction.

Variables that need to be prospectively registered and available:

1. Lesion biology data* - Invasive cancer (Y/N)

   - Pure DCIS (Y/N)

   - Tumour type (1: Invasive Ductal Carcinoma, Non-specific type (IDC-NST) , 2: Invasive Lobular Carcinoma (ILC), 3: Mixed ductolobular carcinoma, 4: Other invasive subtypes, 5: Ductal Carcinoma In Situ (DCIS)

   - Nuclear Grade

   - Estrogen Receptor (ER)
   * Progesterone Receptor (PR)
   * Human Epidermal growth factor Receptor type 2 (HER2 status or erbb-2 status)
   * Ki67% (optional)
   * Any gene signature test (optional)
   * Tumour Infiltrating Lymphocytes (TIL) and Programmed Death Ligand-1 (PDL-1), provided that their report becomes standard of care. (optional)
   * For surgery following neoadjuvant, Residual Cancer Burden (optional) *: Can be replicated from postoperative data in non-discordant cases.
2. Baseline Radiologic Assessment

   - Tumor size (d: maximum diameter in cm). If there is a discrepancy, then the size of the modality (Mammogram, US, MRI) on which the decision is made needs to be registered

   - Localization in the chest (Clock axis, cm from NAC); to be divided into the following categories during harmonization (Upper Outer Quadrant, Junction between Upper and Lower Outer Quadrant, Lower outer quadrant, Junction between Lower Outer and Lower Inner Quadrant, Lower Inner Quadrant, Junction between Lower and Upper Inner Quadrant, Upper Inner Quadrant, Junction between Inner and Outer Upper Quadrant, Retroareolar, Multiple site ipsilateral cancers (previously described as multifocal or multicentric)

   - Tumor size (max size) and Optimal Resection Volume (ORV = 4 / 3π (d / 2 + 1)3, d: maximum diameter in cm.

   - Calculated Resection Ratio: CRR = ORV / BrV, where BrV stands for Breast Volume (see below).
3. Baseline patient assessment:

   * Age at operation
   * Comorbidities (Charlson Comorbidity Index)
   * Smoking
   * Diabetes Mellitus with end-organ damage
   * Neoadjuvant therapy
   * Body mass index (BMI)
   * Ptosis (to be assessed according to the "Regnault" classification, as follows: 1) first degree: nipple at the level of the infra-mammary fold. 2) second degree: nipple below the level of the infra-mammary fold but above the level of the most dependent (inferior) part of the breast contour and 3) third degree: nipple below the level of the infra-mammary fold and sitting at the most dependent, inferior part of the breast contour
   * Breast volume estimate

Acceptable alternatives:

i) "Longo" Formula ii) Breast Cups iii) Bra cup size, if available literature on the conversion of cup size to volume is available) All measurements will be cross-validated by review of preoperative mammograms and calculation of the volume with either the "Kalbhen" or the "Katariya" formulae.

(Kalbhen formula: BrV = 0.784x H x W x C, where H: is anteroposterior distance, W: is mediolateral distance, C: mammographic compression, all in centimeters on the craniocaudal projection of the mammogram ("CC image"), Katariya formula: BrV=π/12*W2*H on the CC image).

* Tumor size (max size) and Optimal Resection Volume (ORV = 4 / 3π (d / 2 + 1) 3, d: maximum diameter in cm.
* Calculated Resection Ratio: CRR = ORV / BrV.
* The rationale behind the recommendation:

To avoid mastectomy; to avoid volume displacement with asymmetry or the need for contralateral symmetrization; to avoid wide local excision with poor cosmetic outcomes.

This assessment will be cross-validated by the team of local PIs

d. Intraoperative data

- Type of volume replacement. The following alternatives are available: Lateral Intercostal Artery Perforator (LICAP), Lateral Thoracic Artery Perforator (LTAP), Lateral Hybrid (combination of LTAP and LICAP), Lateral advancement flap (LAF), Mini Latissimus Dorsi (Muscle sparing), TDAP, Medial or Anterior Intercostal Artery Perforator (MICAP/AICAP), Abdominal Advancement Flap (AAF).

* Single perforator-based flap
* Technique of placement (trapdoor, pendulum, propeller) (optional)
* Tumour localization technique regardless of type (ink, coal, guidewire, seed). Type of localization to be reported
* Axillary procedure (None, SLND, Axillary biopsy, TAD, ALND)
* Specimen weight (in grams, gr)
* Specimen shape, dimensions, and volume (Actual Resection Volume, ARV). The proposed methods are weight/0.958 or volumetry by registration of shape and dimensions.

Specimens are either rectangular and the volume is provided by the formula "V= h x w x l" or elliptical and the volume is provided by the formula "V= 4/3 x (h/2) x (w/2) x (l/2)= 0.654 x h x w x l", where "h": height (cm), "w": width (cm), and "l": length (cm) of the specimen.

* Operative time (min)
* Perioperative antibiotics (Y/N)
* Extended antibiotic administration (Y/N).
* Use of drains
* Day surgery (Y/N)
* Length of stay (days)

  e. Postoperative data
* e.1 Pathology report
* Invasive cancer (Y/N)
* Pure DCIS (Y/N)
* Tumour type (1: IDC, 2: ILC, 3: Mixed, 4: Other invasive, 5: DCIS, 6: Unknown)
* Nuclear Grade (1,2,3)
* Estrogen Receptor (ER) (%)
* Progesterone Receptor (PR) (%)
* HER2 (positive, negative)
* Ki67% -- Tumour Infiltrating Lymphocytes (TIL) and Programmed Death Ligand-1 (PDL-1), provided that their report becomes standard of care.
* Radical excision (Y/N), internationally defined as no "tumour-on-ink" for IBC and 2mm for pure DCIS. National variations in practice will be accepted if they modify the decision-making
* Need for reoperation for complication or margin control (Y/N)
* Type of reoperation (Re-excision, Mastectomy).
* Actual Resection Ratio (ARR), defined as (Specimen volume/Breast volume)
* Number of lymph nodes retrieved (Sentinel and total) (optional)
* Number of lymph nodes with metastases. (to define pN status)
* Type of metastasis (optional)
* e2 Complications at 28 days. Report type.
* Fat necrosis: report Grade according to scale from Lovey et al as follows:

  0 No fat necrosis
  1. Asymptomatic fat necrosis (only radiologic and/ or cytologic ﬁndings)
  2. Symptomatic fat necrosis not requiring medication (palpable mass with or without mild pain)
  3. Symptomatic fat necrosis requiring medication (palpable mass with signiﬁcant pain)
  4. Symptomatic fat necrosis requiring surgical intervention
* Alleged infection (clinical diagnosis)
* Infection (Verified with culture)
* Bleeding
* Symptomatic seroma requiring intervention
* Reporting of complications per the "Clavien Dindo" (CD) classification and Comprehensive Complication Index 2.0 (CCI 2.0) score.
* e3 Type of (Neo)Adjuvant Systemic therapy (None, Chemotherapy, Endocrine Therapy, Monoclonal antibodies, CDK 4-6 inhibitors or other)
* e4 Type of Adjuvant Radiotherapy (None, whole breast irradiation, reduced dose whole breast irradiation, partial breast irradiation plus minus nodal/regional irradiation) f. Patient Reported Outcomes (Optional) Questionnaires accepted

EORTC QLQ-c-30 BreastQ preoperative and postoperative modules Diseases of the Arm, Shoulder and Hand (DASH) score

g. Health-economy outcomes

h. Long-term follow-up Ipsilateral Local recurrence Ipsilateral Locoregional recurrence Distant Recurrence Breast Cancer-Specific Survival Overall Survival (All in months).

ELIGIBILITY:
Inclusion Criteria:

1. Female aged above 18 years.
2. Signed and dated written informed consent before the start of specific protocol procedures; oral consent for the participants of the quality control retrospective cohort study before accepting to partake a telephone interview.
3. Patients with invasive breast cancer (IBC) or ductal cancer in situ (DCIS) or unclear lesions mandating surgical excision or benign lesions amenable for surgical resection with BCS.
4. ECOG performance status 0-2.

Exclusion Criteria

1. Life expectancy of less than 6 months
2. Non candidate for breast conservation
3. Inability to understand given information and give informed consent or undergo study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As discussed above
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Avoidance of mastectomy | 3 months
  Percenteage of patients not amenable to standard wide local excision following a standardized assessment, that are operated with oncoplastic breast conservation resulting in negative margins and avoid mastectomy.
Re-excision rates | 3 months
  Percenteage of patients not amenable to standard wide local excision following a standardized assessment, that undergo breast conservation, but require re-excision of margins without conversion to mastectomy as a final result.
Patient reported outcomes, European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (QLQ-C30) | Baseline, postoperative (6, 12, 24 months)
  The European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (QLQ-C30) is a validated 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients. It assesses both quality of life domains and symptom domains in a scale score ranging from 0 to 100. For the quality of life domains, higher scores denote higher satisfaction or higher quality of life. For symptom scales, higher score denotes more severe symptoms. In the Summary Score of the Questionnaire, higher values denote higher quality of life
Patient reported outcomes, BreastQ module for Satisfaction with Breasts | Baseline, postoperative (6, 12, 24 months)
  The BREAST-Q questionnaire is developed especially for breast cancer patients undergoing breast surgery. Independent modules are available for the different surgical interventions (e.g., mastectomy, reconstruction, augmentation). The BREAST-Q questionnaire has been validated and serves as of a standardized measurement instrument. The Satisfaction with Breasts module is summarized in a score ranging from 0 to 100, with higher scores denoting higher satisfaction
Patient reported outcomes, BreastQ module for Physical Wellbeing: Chest | Baseline, postoperative (6, 12, 24 months)
  The BREAST-Q questionnaire is developed especially for breast cancer patients undergoing breast surgery. Independent modules are available for the different surgical interventions (e.g., mastectomy, reconstruction, augmentation). The BREAST-Q questionnaire has been validated and serves as of a standardized measurement instrument. The Physical Wellbeing: Chest module is summarized in a score ranging from 0 to 100, with higher scores denoting higher wellbeing

SECONDARY OUTCOMES:
Postoperative Complications | 6 weeks or up to 3 months if no other adjuvant oncologic treatment has been employed
  Postoperative complications, reported descriptively, per the modified Clavien Dindo classification and the Comprehensive Complication Index 2.0 (CCI 2.0)
Operative time | At surgery
  Operative time in minutes
Length of stay | Perioperative
  Number of days of inpatient care
Profile of mastectomy candidates | Preoperative
  Characteristics of patients that require mastectomy per surgeon assessment
Procedure-related costs | Postoperative
  Costs related with each surgical procedure
Local Recurrence Free Survival | Up to 10 years
  Time from Surgery to ipsilateral local recurrence (in situ or invasive)
Locoregional Recurrence Free Survival | Up to 10 years
  Time from Surgery to ipsilateral locoregional recurrence (in situ or invasive)
Disease Free Survival | Up to 10 years
  Time from Surgery to any recurrence
Breast Cancer Specific Survival | Up to 10 years
  Time from surgery to breast cancer related death
Overall Survival | Up to 10 years
  Time from surgery to death from any cause

OTHER OUTCOMES:
Type of axillary surgery | At surgery
  Type of axillary procedure performed at the time of breast surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Karakatsanis, MD, PhD, Principal Investigator — Uppsala University
Locations (3):
- Westmead Breast Cancer Institute, Sydney, Australia
- Uppsala University Hospital, Uppsala, Sweden
- Royal Marsden Hospital, London, United Kingdom